CLINICAL TRIAL: NCT02753205
Title: Effect of Dexmedetomidine on Optic Nerve Sheath Diameter During Laparoscopic Anterior Resection
Brief Title: Dexmedetomidine on Optic Nerve Sheath Diameter
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCIRB2016-058
Record Dates: First submitted 2016-04-14; First posted 2016-04-27 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Intracranial Hypertension
MeSH Terms: conditions — Intracranial Hypertension | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Experimental): Infusion of normal saline
  Interventions: Drug: normal saline
- Dexmedetomidine (Active Comparator): infusion of dexmedetomidine 0.5ug/kg/h for 10 min and after that, infusion of dexmedetomidine 0.4ug/kg/h until the end of surgery
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — infusion of dexmedetomidine 0.5ug/kg/h for 10 min and after that, infusion of dexmedetomidine 0.4ug/kg/h until the end of surgery
  Other Names: dex
  Arms: Dexmedetomidine
Drug: normal saline — infusion of normal saline
  Other Names: NS
  Arms: Control

SUMMARY:
Dexmedetomidine, might attenuate the sympathetic activation and contribute to stable hemodynamics. The investigator hypothesized that continuous infusion of dexmedetomidine during laparoscopic lower abdominal surgery, might help to attenuate the increment of intracranial pressure and the investigator would observe the optic nerve sheath diameter using ultrasonography.

DETAILED DESCRIPTION:
Laparoscopic lower abdominal surgery requires the Trendelenburg position with pneumoperitoneum for a prolonged time, but this can cause significant increase in intracranial pressure. Dexmedetomidine, a selective alpha2 receptor agonist might attenuate the sympathetic activation and contribute to stable hemodynamics. The investigator hypothesized that continuous infusion of dexmedetomidine during laparoscopic lower abdominal surgery, might help to attenuate the increment of intracranial pressure and the investigator would observe the optic nerve sheath diameter using ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of colorectal cancer
* planed for laparoscopic low anterior resection

Exclusion Criteria:

* morbid obesity (body mass index > 30 kg.m-2)
* history of cerebrovascular disease
* history of respiratory disease
* uncontrolled cardiovascular disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | Change from Baseline optic nerve sheath diameter at pneumoperitoneum 30 min
  mm

SECONDARY OUTCOMES:
Respiratory and mean arterial pressure | Change from Baseline Respiratory and mean arterial pressure at pneumoperitoneum 30 min
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, Study Chair — Gachon Universtiy Gil Medical Center

IPD SHARING:
Plan to Share IPD: No